CLINICAL TRIAL: NCT04438057
Title: Evaluating the Efficacy of Convalescent Plasma in Symptomatic Outpatients Infected With COVID-19
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Metro Infectious Disease Consultants (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MIDC-CCP
Record Dates: First submitted 2020-06-17; First posted 2020-06-18 (Actual); Last update posted 2022-04-06 (Actual); Status verified 2022-04

CONDITIONS: COVID-19
Keywords: convalescent plasma
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Intervention Model Description: Outpatient open label randomized study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Standard of Care (No Intervention): Patient will receive standard of care therapy.
- Treatment Arm (Active Comparator): Patient will receive convalescent plasma
  Interventions: Biological: CCP

INTERVENTIONS:
Biological: CCP — Randomized open label study to receive 2:1 CCP to standard of care
  Other Names: convalescent plasma
  Arms: Treatment Arm

SUMMARY:
This study will provide investigational convalescent plasma for patients infected with the SARS-CoV-2 with mild to moderate symptoms who meet inclusion criteria as judged by physician evaluation.

DETAILED DESCRIPTION:
This study will provide investigational convalescent plasma for patients infected with the SARS-CoV-2 with mild to moderate symptoms who meet inclusion criteria as judged by physician evaluation.

Following patient enrollment into the study, completion of informed consent and randomization, the patient will receive one unit of convalescent COVID plasma or standard of care. The plasma will be infused in an outpatient infusion center by highly trained and experienced staff. Vitalant will be providing the plasma as per their normal screening and distribution protocols. Patients will be monitored for safety during the infusion and per protocol following the infusion for a period of 28 days. Primary efficacy and safety endpoints will be statistically analyzed and compared between the two groups.

ELIGIBILITY:
Inclusion Criteria:

* Laboratory confirmed diagnosis of infection with SARS-CoV-2
* Symptoms of COVID -19 - cough, fever, sore throat, SOB, anosmia, diarrhea, myalgia
* Symptoms less than 14 days
* ID Physician determination that the patient does not need hospitalization
* O2 saturation of >93%
* Informed consent provided by the patient or healthcare proxy
* Age ≥ 18 years
* Ambulatory Outpatient when informed consent obtained and study drug is administered

Exclusion Criteria:

* Age < 18 y/o
* Patients currently receiving intravenous immunoglobulin
* Hypercoagulable state - neoplasia, Collagen vascular disease, Myelodysplastic syndrome, chronic anticoagulation treatment, etc.
* Need to be hospitalized
* O2 sat < 93%
* D-Dimer > 2x normal
* Chronic oxygen therapy
* Renal insufficiency with Creatinine clearance < 30
* Long term care or assisted living facility resident
* Ongoing usage of hydroxychloroquine for any indication
* History of blood or plasma transfusion related complications
* Enrollment into any other investigational drug or device study within the previous 30 days
* Any drug, chemical or alcohol dependency as determined by the investigator through history that may affect study procedures and follow up
* Pregnant or breast feeding
* Any acute or chronic medical comorbidity, psychiatric, social or other circumstance that, in the opinion of the investigator, may interfere with study compliance, completion, or accurate assessment of the study outcomes/safety
* Admitted to or expected to be admitted to a medical facility

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 103 (Actual)
Dates: Start 2020-08-12 (Actual); Primary Completion 2020-08-12 (Actual); Study Completion 2021-08-12 (Actual)

PRIMARY OUTCOMES:
Time to Resolution of Symptoms | 28 days
  a. Time to resolution of symptoms will be defined as time from randomization (day 0) to a successful outcome. c. A successful outcome is defined as symptom improvement of 3 numbers or down to zero on the memory aid for all symptoms noted.
SAEs within 24 hours of plasma infusion | 28 days

SECONDARY OUTCOMES:
Decrease in Inflammatory Markers | 28 days
  A 50% decrease at day 28 in C-Reactive Protein (mg/mL)
Decrease in Inflammatory Markers | 28 days
  A 50% decrease at day 28 in D-Dimer (ng/mL)
Decrease in Inflammatory Markers | 28 days
  A 50% decrease at day 28 in Ferritin (ng/mL)
Decrease in Inflammatory Markers | 28 days
  A 50% decrease at day 28 in Lactate Dehydrogenase (U/L)
Hospitalization within 28 days | 28 days

CONTACTS AND LOCATIONS:
Locations (1):
- Metro Infectious Disease Consultants, Burr Ridge, Illinois, United States

IPD SHARING:
Plan to Share IPD: No